CLINICAL TRIAL: NCT01499472
Title: ESWT Treatment of Diabetic Foot VS. Standard Care Trial
Brief Title: Comparing the Expected Benefit of Extra-corporeal-shockwave Therapy (ESWT) Treatment to Standard Care in Treating Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ofer Elishuv, Doctor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ofer02-HMO-CTIL
Record Dates: First submitted 2011-09-04; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Extracorporeal Shockwave Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- shock wave therapy, shortened wound healing time (Active Comparator)
  Interventions: Device: shock wave therapy; Device: dermagold shockwave
- normal wound care (Other): standard of care intervention
  Interventions: Procedure: standard of care

INTERVENTIONS:
Device: shock wave therapy — shock wave therapy given in accordance to wound assessment every 2 weeks for 4 treatments.
  Arms: shock wave therapy, shortened wound healing time
Device: dermagold shockwave — shock wave therapy given in accordance to wound assessment every 2 weeks for 4 treatments.
  Arms: shock wave therapy, shortened wound healing time
Procedure: standard of care — regular care including debridement and bandaging.
  Arms: normal wound care

SUMMARY:
The purpose of this study is to determine if Extra-corporeal-shockwave Therapy (ESWT) added to standard of care wound therapy significantly improves time to complete wound healing in diabetic foot wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent.
2. Diagnosed with Diabetes.
3. An Active Diabetic Ulcer larger than 5 cm2
4. Sufficient limb perfusion.(e.g no compartment syndrome ankle Brachial Index (ABI)>=0.5

Exclusion Criteria:

1. Pregnancy.
2. The patient is under another research protocol.
3. One of the following:

   A. ABI<0.5 C.Significant Arterial-Venous injury. D. Lymphedema.
4. The patient underwent Chemotherapy or Radiotherapy 60 days or less prior to recruitment date.
5. Sufficient Noncompliant.
6. Sickle Cell Anemia, HIV, Immunodeficiency, HgB Anemia, DVT, Chronic Renal Failure, Systemic use of Steroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
healed ulcer | 6 months